CLINICAL TRIAL: NCT00179998
Title: Efficacy of Pulmozyme in Infants and Young Children With Cystic Fibrosis
Brief Title: Effectiveness of Pulmozyme in Infants With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z2910s
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Infants; Children; Pulmozyme; Pulmonary function; Computed tomography
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant Human DNase (Pulmozyme) then Placebo (Active Comparator): once daily nebulized rhDNAse
  Interventions: Drug: Recombinant Human DNase (Pulmozyme); Drug: Placebos
- Placebo (Nebulized Saline) then rhDNase (Placebo Comparator): once daily nebulized vehicle
  Interventions: Drug: Recombinant Human DNase (Pulmozyme); Drug: Placebos

INTERVENTIONS:
Drug: Recombinant Human DNase (Pulmozyme) — 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
  Other Names: Pulmozyme
Drug: Placebos — 2.5 ml sterile solution (8.77 mg/ml sodium chloride, 0.15 mg/ml calcium chloride, pH 7.0 +/- 2.0) delivered daily by nebulization for 6 months, either preceding or following 6 months of Pulmozyme depending on randomization of the subject

SUMMARY:
This is a study to find out whether Pulmozyme is effective for clearing mucus from the airways of children with cystic fibrosis less than 3 ½ years of age.

DETAILED DESCRIPTION:
Pulmozyme is given using a nebulizer and is now widely used in older children and adults with cystic fibrosis. In adults and older children, studies have shown that daily use of Pulmozyme improves lung function and decreases the number of lung infections requiring hospital treatment. Pulmozyme has been approved by the Food and Drug Administration for use in children over 5 years old and adults with cystic fibrosis. Pulmozyme has also been approved by the FDA for use in children with cystic fibrosis less than 5 years old based upon studies showing that it is safe in this age group and that it does get into the airway tubes as well in infants and toddlers as it does in older children and adults. Currently Pulmozyme is not widely used in children with cystic fibrosis younger than 5 years because no study has clearly shown that inhaling Pulmozyme daily improves lung function or improves clearance of mucus from the airway tubes in very young children. This study will measure whether Pulmozyme improves lung function and mucous clearance from the lungs in children with cystic fibrosis less than 3 ½ years of age.

This study will compare Pulmozyme to a placebo. During the study infants and young children with cystic fibrosis will be treated with Pulmozyme for 6 months and placebo for 6 months. The study medicines will be inhaled at home once a day from a nebulizer for a period of one year. Half of the children will be treated with Pulmozyme for the first 6 months of the study and half will receive the placebo. At the 6 month point the group receiving Pulmozyme will be changed to the placebo and the group receiving placebo will be changed to Pulmozyme. The order of the 6 month treatment periods is randomized. This study is blinded. The study doctor and his staff will not know who is receiving Pulmozyme or placebo at any time during the study.

Whether Pulmozyme works will be measured using infant lung function tests and by doing a special 3-D x-ray of the child's chest (a high resolution CT or HRCT) at the beginning of the study, at 6 months and at 12 month after starting study. The study will not change the regular clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age < 30 months
* Diagnosis of CF based on clinical features consistent with CF as well as 1 of the 2 following criteria: a) two sweat chlorides >60 mEq/L (by quantitative pilocarpine iontophoresis), b) genotype with 2 identifiable mutations consistent with CF.
* Informed consent by parent or legal guardian

Exclusion Criteria:

* Previous treatment with Pulmozyme
* Hospitalization or treatment with IV antibiotics with 14 days of initial study visit
* Acute intercurrent respiratory infection, defined as any of the following symptoms within the preceding 48 hours: 1) fever > 38 degrees C, 2) new onset of coryza or other upper respiratory symptoms, 3) increase in cough, wheezing, or respiratory rate
* History of adverse reaction to sedation
* Oxyhemoglobin saturation <90% on room air
* Severe upper airway obstruction as determined by site PI (severe laryngomalacia, markedly enlarged tonsils, significant snoring, diagnosed obstructive sleep apnea)
* Hemodynamically significant congenital heart disease or diagnosed arrhythmias
* History of hemoptysis
* History of previous pulmonary air leak (pneumothorax)
* Diagnosed seizure disorder necessitating current anticonvulsive therapy. A history of febrile seizures is not an exclusion criterion.
* Use of Investigational drug(s) within 60 days or 5 half-lives of enrollment in this study.
* Known allergy to Chinese Hamster Ovary-derived biological products or any component of the placebo or active drug formulations.

Ages: 1 Month to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Castile, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - rhDNase Then Placebo: once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
- 2 - Placebo Then rhDNase: once daily nebulized vehicle
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
Period: Initial Period - 6 Months
Arm/Group | 1 - rhDNase Then Placebo | 2 - Placebo Then rhDNase
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Crossover Period - 6 Months
Arm/Group | 1 - rhDNase Then Placebo | 2 - Placebo Then rhDNase
Started | 12 | 12
Completed | 12 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Nebulized rhDNAse Then Placebo: once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months then 3 ml diluent placebo delivered by nebulization given daily for 6 months
- Placebo Then Nebulized rhDNAse: once daily nebulized vehicle
  Recombinant Human DNase (Pulmozyme): Comparison of 3 ml diluent placebo delivered by nebulization given daily for 6 months then 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months
- Total: Total of all reporting groups
Arm/Group | Nebulized rhDNAse Then Placebo | Placebo Then Nebulized rhDNAse | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 23.3 (11.9) | 48.3 (36.7) | 41.8 (31.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Chest CT (High Resolution Computed Tomography (HRCT) Score)
Description: Change in Total HRCT Score from initiation of intervention to 6 months
  Modified Maffessanti HRCT Scoring System
  Airways
  1. Bronchial Wall Thickening:1 = mild, 2 = moderate, 3 = severe
  2. Bronchiectasis:1 = mild, 2 = moderate, 3 = severe
  3. Axial extent of 1 or 2: 1 = central/middle, 2 = also periphery
  4. Regional extent of 1 or 2: x 1 if < 50 %, x 2 if > 50 %
  5. Gas trapping score:0 if 1 sub-segment, 1 if < 25 %, 2 if 25 - 50 %, 3 if 50 - 75 %, 4 if > 75 % Multiply (# 1 + # 2 + # 3) by # 4 then add # 5
  Parenchyma
  1. Airspace disease: 0 = none, 1 = present
  2. Ground glass opacity: 0 = none, 1 = present
  3. Mucous Plugging: 0 = none, 1 = present
  Total Score = Airway + Parenchymal Scores for RUL, LUL, RLL, and LLL Sections. The Total Score ranges from 12 to 92, with higher scores indicating greater impairment.
  Maximum Score = 4 x 23 = 92
Time Frame: 6 months
Population: Subjects will include children with CF < 30 months old and never treated with Pulmozyme. Patients available for recruitment will include 12 newly diagnosed children <30 months old from Nationwide Children's Hospital and 4 from Dayton Children's.
Measure: Mean (Standard Deviation); unit: Score points
Groups:
- Nebulized rhDNAse: once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
- Nebulized Saline: once daily nebulized vehicle
Arm/Group | Nebulized rhDNAse | Nebulized Saline
Number analyzed (Participants) | 12 | 12
Score points | 3.7 (21.1) | 6.1 (9.5)

2. Primary Outcome: Infant Pulmonary Function Tests (FEV0.5)
Description: Change in FEV0.5 from initiation of intervention to 6 months
Time Frame: 6 months
Population: Children < 30 months of age with cystic fibrosis who were given either the study drug followed by the placebo or given placebo followed by study drug. Data is not available for the second period, as the PI has retired and is no longer associated with NCH.
Measure: Mean (Standard Deviation); unit: z score
Groups:
- Nebulized rhDNAse Then Placebo: once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
- Placebo (Nebulized Saline) Then rhDNAse: Once daily 3 ml diluent delivered by nebulization given daily for 6 months followed by 2.5 mg rhDNAse in 3 ml diluent delivered by nebulization given daily for 6 months
Arm/Group | Nebulized rhDNAse Then Placebo | Placebo (Nebulized Saline) Then rhDNAse
Number analyzed (Participants) | 12 | 12
z score | -0.1 (1.1) | -0.2 (1.0)

3. Secondary Outcome: Antibiotic Treatment Days
Description: Total number of days treated with IV, oral or nebulized antibiotics over 6 initial month interval
Time Frame: per 6 month interval
Population: Subjects included children < 30 months of age who were newly diagnosed with Cystic Fibrosis. Subjects were recruited from Nationwide Children's (AKA Columbus Children's) and Dayton Children's Hospitals.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Nebulized rhDNAse Then Placebo: once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent. IPFTs and CV-HRCT will be performed at that time. These subjects will then receive the placebo (Normal saline) delivered by nebulization given daily for 6 months. IPFT and CV-HRCTs will be performed again at 1 year.
- Placebo (Nebulized Saline) Then rhDNAse: Those placed in the placebo arm with receive nebulized normal saline daily for 6 months. Following evaluation by IPFT and CV-HRCT, these subjects will receive the study drug daily for 6 months by the same delivery method. IPFT and CT-HRCTs will be performed again at 1 year.
Arm/Group | Nebulized rhDNAse Then Placebo | Placebo (Nebulized Saline) Then rhDNAse
Number analyzed (Participants) | 12 | 12
days | 31.7 (24.5) | 36.3 (20.1)

ADVERSE EVENTS:
Time Frame: 6 months for each intervention
Description: Safety population included all participants who received either the study drug or placebo
Groups:
- Nebulized rhDNAse Then Placebo(Nebulized Saline): once daily nebulized rhDNAse
  Recombinant Human DNase (Pulmozyme): Comparison of 2.5 mg in 3 ml diluent delivered by nebulization given daily for 6 months with 3 ml diluent placebo delivered by nebulization given daily for 6 months
  Data is unavailable for the second period. The PI has retired and is no longer associated with the institution.
- Placebo (Nebulized Saline) Then rhDNAse: Once daily nebulized saline daily for 6 months, followed by Recombinant Human DNase (Pulmozyme) in 3 ml diluent daily for 6 months
  Data is unavailable for the second period. The PI has retired and is no longer associated with the institution.
Arm/Group | Nebulized rhDNAse Then Placebo(Nebulized Saline) | Placebo (Nebulized Saline) Then rhDNAse
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulized rhDNAse Then Placebo(Nebulized Saline) (N=12) | Placebo (Nebulized Saline) Then rhDNAse (N=12)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — child hospitalized for treatment of wheezing 4 months after starting Nebulized rhDNAse. Data is not available for the second period.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulized rhDNAse Then Placebo(Nebulized Saline) (N=12) | Placebo (Nebulized Saline) Then rhDNAse (N=12)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11) — Cough reported at any monthly assessment over 6 month study interval

LIMITATIONS AND CAVEATS:
Dr. Castile is retired and no longer is associated with Nationwide Children's Hospital and no one associated with the trial works at NCH any longer. We are unable to further update this study in clinicaltrials.gov.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No